CLINICAL TRIAL: NCT07235293
Title: A Randomized, Open-label, Phase 2b Study to Compare the Efficacy of DSP107 in Combination With Atezolizumab Versus Fruquintinib in Patients With Advanced Microsatellite Stable Colorectal Cancer
Brief Title: A Study to Test DSP107 in Combination With Atezolizumab in Comparison With Fruquintinib as a New Treatment for Colorectal Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kahr Bio Australia Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Kahr Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSP107_003
Record Dates: First submitted 2025-11-03; First posted 2025-11-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DSP107 in combination with Atezolizumab (Experimental): DSP107 10 mg/kg IV on Days 1, 8, and 15 of each 28-day cycle. Atezolizumab 1680 mg IV on Day 1 of each 28-day cycle.
  Interventions: Drug: DSP107 + Atezolizumab
- Fruquintinib (Active Comparator): Participants will receive fruquintinib orally in 28-day cycles, for up to 24 cycles (96 weeks), or until disease progression, unacceptable toxicity, or study withdrawal.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: DSP107 + Atezolizumab — DSP107 infusion begins ~30 (±10) minutes after completion of atezolizumab infusion on Day 1.
  Arms: DSP107 in combination with Atezolizumab
Drug: Fruquintinib — 5 mg orally, once daily (with or without food), on Days 1-21 of each 28-day cycle, followed by 7 days off.
  Arms: Fruquintinib

SUMMARY:
This clinical study is testing whether a new combination of medicines (DSP107 and atezolizumab) is more effective and safer than an existing treatment (fruquintinib) for people with advanced colorectal cancer that is microsatellite stable (MSS). Participants will be randomly assigned to receive one of the two treatments, and researchers will monitor how well the cancer responds, how safe the treatments are, and how the body processes them. The study hopes to show that the new combination can improve outcomes for patients with this type of colorectal cancer.

DETAILED DESCRIPTION:
This Phase 2b, randomized, open-label, multicenter study will enroll participants with advanced MSS or mismatch repair-proficient (pMMR) colorectal cancer who have progressed on, or shown intolerance to, standard therapies, including fluoropyrimidine, irinotecan, oxaliplatin, trifluridine/tipiracil (Lonsurf), bevacizumab, and epidermal growth factor receptor (EGFR) inhibitors if RAS wild-type. Participants with BRAF V600E mutation, HER2 amplification/overexpression, KRAS G12C mutation, RET fusion, or NTRK fusion may also have received one prior targeted therapy. Prior treatment with fruquintinib or regorafenib is not allowed.

Participants will be randomized 1:1 into two arms:

Group A (Experimental): DSP107 10 mg/kg intravenously on Days 1, 8, and 15 of each 28-day cycle, administered after atezolizumab 1680 mg IV on Day 1 of each cycle. DSP107 infusion may be shortened after initial tolerance. Atezolizumab infusion may be shortened from 60 to 30 minutes if well tolerated.

Group B (Active Comparator): Fruquintinib 5 mg orally once daily on Days 1-21 of each 28-day cycle, with dosing diaries maintained by participants.

Total duration of study participation for each participant will vary based on factors including treatment tolerability, disease progression and other study discontinuation criteria.

Study duration for participants will include at least:

* Screening Period of up to 28 days
* Treatment Period of up to 24 cycles of 28 days
* Safety Follow-up Period of up to 90 days* from the last dose of IP or active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥ 18 years of age with a life expectancy of > 3 months.
2. Participants with histologically confirmed, inoperable, MSS and/or pMMR CRC which has progressed to, or is intolerant to, specified therapies (and has received prior treatment with no more than 3 lines of therapy).

   Note: Lines of therapy are defined by disease progression between therapies. Participants who discontinue their prior regimen due to toxicity (in the absence of disease recurrence/progression) will also have their prior therapy count as one prior regimen.
3. Measurable disease per RECIST v1.1.

Exclusion Criteria:

1. Central nervous system (CNS) metastases unless stable 2 months post definitive therapy with steroids.
2. Unresolved AEs of Grade 2 or higher from prior anticancer therapy.
3. Past or current history of autoimmune disease or immune deficiency.
4. History of other malignancy within 3 years of first study treatment cycle.
5. Current or recent treatment with certain therapies including specified anticancer treatments, modulators of CYP3A4 and immunomodulating therapies (prior treatment with CPIs is not exclusory).
6. Known allergy or hypersensitivity to any of the test compounds, materials, or contraindication to test product.
7. Clinically significant abnormal laboratory safety tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
To determine Median overall survival (mOS) in participants treated with the combination of DSP107 and atezolizumab versus fruquintinib. | From Day 1 until date of death from any cause assessed up to 2 years
  Median Overall Survival (mOS) will be estimated using Kaplan-Meier methodology as the median time from the start of study treatment to the last known date a participant was alive. Censoring rules will be applied for participants without an event at the time of analysis, and 95% confidence intervals for mOS will be provided.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From Screening to Follow-up (30 to 90 Days Post IP)
  Safety and tolerability of DSP107 + atezolizumab versus fruquintinib, assessed by incidence and severity of AEs per CTCAE v5.0 (including SAEs and AESIs).
Changes in 12-lead ECG parameters | From Baseline through to end of treatment visit, an average of 6 months
  Safety assessment based on changes from baseline in ECG intervals (PR, QRS, QT, QTc) and heart rate.
Change in Overall Survival (OS) | From randomization through study participation, with survival follow-up for up to 5 years in the DSP107_SFU study.
  On completion of the safety follow-up, participants will be requested to enroll on protocol DSP107_SFU ("Observational, long-term survival follow-up study of participants previously treated in DSP107 interventional study") to allow determination of overall survival. After receiving written informed consent, all participants will be followed for up to 5 years on the DSP107_SFU study.
Change from Baseline in Quality of Life (QoL) | From Baseline through to end of treatment visit, an average of 6 months
  Evaluation of the effect of treatment on quality of life (QoL) using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Change from Baseline in Systolic and Diastolic Blood Pressure | From Baseline through to end of treatment visit, an average of 6 months
  Mean change from baseline in blood pressure (mmHg).
Change from Baseline in Pulse Rate | From Baseline through to end of treatment visit, an average of 6 months
  Mean change from baseline in heart rate (beats per minute).
To evaluate the immunogenicity of DSP107 when administered in combination with atezolizumab. | From Baseline through to end of treatment visit, an average of 6 months
  Immunogenicity will be assessed by measurement of anti-drug antibodies (ADAs) to DSP107 in serum samples collected at specified time points.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - University of Colarodo Cancer Center, Aurora, Colorado
  - Mayo Clinic, Florida City, Florida
  - Duke Cancer Institute - Duke Cancer Center, Durham, North Carolina
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Texas City, Texas
- Australia (11):
  - The Queen Elizabeth Hospital, Woodville, Adelaide
  - Chris O'brien Lifehouse, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre, South Brisbane, Queensland
  - Flinders Medical Centre SA, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Footscray Hospital - Western Health, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Sunshine Hospital - Western Health, Saint Albans, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No